CLINICAL TRIAL: NCT00616876
Title: The Effects of Lactulose Supplementation to Enteral Feedings in Premature Infants - A Pilot Study
Brief Title: Lactulose Supplementation in Premature Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Arieh Riskin MD, Bnai Zion Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: BZ-23/04; LacPre18
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Necrotizing Enterocolitis; Sepsis
Keywords: lactulose; prebiotic; premature infant; enteral feeding; stools; lactobacillus; nutrition; growth
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis; Premature Birth | interventions — Lactulose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Study group will receive 1% lactulose in all their feeds (human milk or preterm formula)
  Interventions: Drug: Lactulose
- 2 (Placebo Comparator): Control group will receive 1% dextrose placebo in all their feeds (human milk or preterm formula).
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Drug: Lactulose — Babies in the study group received lactulose in a dose of 1% in their entire mother's breast milk or preterm formula feeds (1 gram per 100 ml feeds, based on the daily volume of feeds, and evenly distributed between all the feeds for the entire duration of their hospital stay). 67% lactulose in the original preparation (Laevolac, Fresenius Kabi, Austria) was diluted by distilled water to 33.5% preparation in the pharmacy in strict sterile conditions under hood. Just before feeding the nurses added the required volume of this 33.5% lactulose solution to the ordered volume of feed to generate a final concentration of 1% lactulose in each feed.
  Arms: 1
Dietary Supplement: Dextrose — Babies in the control groups were given equal volumes of the comparable placebo in all their preterm formula feeds at final concentration of 1% dextrose. The 33.5% dextrose placebo solution was prepared by dissolving dextrose (Dextrose Pulv. USP.24/BP, Roquette Frores 6280, Lestrem, France) in distilled water under heat to the point of near boiling under the same strict sterile conditions in the pharmacy. This gave a placebo solution that looked similar in color, odor and liquidity to the study solution of 33.5% lactulose. Dark bottles were used to further blind the medical team as to what solution was the baby given.
  Arms: 2

SUMMARY:
A pilot study to test the safety of use of lactulose in preterm infants and to preliminary assess the hypothesis that lactulose would support the early growth of Lactobacilli in the stools of premature infants and possibly would also improve nutritional status and decrease NEC and late-onset sepsis.

DETAILED DESCRIPTION:
Prospective, double-blind, placebo-controlled single center pilot study in 23-34 weeks gestation premature infants. Study group will receive 1% lactulose, while control group will receive 1% dextrose placebo in all their feeds (human milk or preterm formula). Clinical parameters will be followed. Stool samples will be sent for culture.

ELIGIBILITY:
Inclusion Criteria:

Premature infants were recruited based on the following criteria:

* 23-34 weeks' gestation (as determined by a combination of maternal dates, early prenatal ultrasonography and postnatal gestational age estimation based on physical and neuromuscular signs (New Ballard Score), as long as there will be gestational age agreement between the 3 methods < 2 weeks);
* Absence of major congenital malformations; and
* Informed consent obtained from parents.

Exclusion Criteria:

* Major congenital malformations and parental refusal.

Ages: 23 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
lactulose would support the early growth of Lactobacilli in the stools of premature infants | 1.5 years

SECONDARY OUTCOMES:
lactulose would also improve nutritional status and decrease NEC and late-onset sepsis in preterm infants | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Riskin, MD, Principal Investigator — Department of Neonatology, Bnai Zion Medical Center; Ron Shaoul, MD, Principal Investigator — Department of Pediatrics, Pediatric Gastroenterology, Bnai Zion Medical Center
Locations (1):
- NICU, Department of Neonatology, Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Background] Rotimi VO, Duerden BI. The development of the bacterial flora in normal neonates. J Med Microbiol. 1981 Feb;14(1):51-62. doi: 10.1099/00222615-14-1-51. PMID 7463467
- [Background] Orrhage K, Nord CE. Factors controlling the bacterial colonization of the intestine in breastfed infants. Acta Paediatr Suppl. 1999 Aug;88(430):47-57. doi: 10.1111/j.1651-2227.1999.tb01300.x. PMID 10569223
- [Background] Benno Y, Sawada K, Mitsuoka T. The intestinal microflora of infants: composition of fecal flora in breast-fed and bottle-fed infants. Microbiol Immunol. 1984;28(9):975-86. doi: 10.1111/j.1348-0421.1984.tb00754.x. PMID 6513816
- [Background] Guarner F, Malagelada JR. Gut flora in health and disease. Lancet. 2003 Feb 8;361(9356):512-9. doi: 10.1016/S0140-6736(03)12489-0. PMID 12583961
- [Background] Vanderhoof JA, Young RJ. Probiotics in pediatrics. Pediatrics. 2002 May;109(5):956-8. doi: 10.1542/peds.109.5.956. No abstract available. PMID 11986461
- [Background] Bennet R, Eriksson M, Nord CE, Zetterstrom R. Fecal bacterial microflora of newborn infants during intensive care management and treatment with five antibiotic regimens. Pediatr Infect Dis. 1986 Sep-Oct;5(5):533-9. doi: 10.1097/00006454-198609000-00009. PMID 3763418
- [Background] Hall MA, Cole CB, Smith SL, Fuller R, Rolles CJ. Factors influencing the presence of faecal lactobacilli in early infancy. Arch Dis Child. 1990 Feb;65(2):185-8. doi: 10.1136/adc.65.2.185. PMID 2317064
- [Background] Sakata H, Yoshioka H, Fujita K. Development of the intestinal flora in very low birth weight infants compared to normal full-term newborns. Eur J Pediatr. 1985 Jul;144(2):186-90. doi: 10.1007/BF00451911. PMID 4043132
- [Background] Caicedo RA, Schanler RJ, Li N, Neu J. The developing intestinal ecosystem: implications for the neonate. Pediatr Res. 2005 Oct;58(4):625-8. doi: 10.1203/01.PDR.0000180533.09295.84. PMID 16189184
- [Background] Gewolb IH, Schwalbe RS, Taciak VL, Harrison TS, Panigrahi P. Stool microflora in extremely low birthweight infants. Arch Dis Child Fetal Neonatal Ed. 1999 May;80(3):F167-73. doi: 10.1136/fn.80.3.f167. PMID 10212075
- [Background] Gaynes RP, Edwards JR, Jarvis WR, Culver DH, Tolson JS, Martone WJ. Nosocomial infections among neonates in high-risk nurseries in the United States. National Nosocomial Infections Surveillance System. Pediatrics. 1996 Sep;98(3 Pt 1):357-61. PMID 8784356
- [Background] Millar M, Wilks M, Costeloe K. Probiotics for preterm infants? Arch Dis Child Fetal Neonatal Ed. 2003 Sep;88(5):F354-8. doi: 10.1136/fn.88.5.f354. PMID 12937036
- [Background] Neu J, Caicedo R. Probiotics: protecting the intestinal ecosystem? J Pediatr. 2005 Aug;147(2):143-6. doi: 10.1016/j.jpeds.2005.05.033. No abstract available. PMID 16126038
- [Background] Dani C, Biadaioli R, Bertini G, Martelli E, Rubaltelli FF. Probiotics feeding in prevention of urinary tract infection, bacterial sepsis and necrotizing enterocolitis in preterm infants. A prospective double-blind study. Biol Neonate. 2002 Aug;82(2):103-8. doi: 10.1159/000063096. PMID 12169832
- [Background] Millar MR, Bacon C, Smith SL, Walker V, Hall MA. Enteral feeding of premature infants with Lactobacillus GG. Arch Dis Child. 1993 Nov;69(5 Spec No):483-7. doi: 10.1136/adc.69.5_spec_no.483. PMID 8285750
- [Background] Agarwal R, Sharma N, Chaudhry R, Deorari A, Paul VK, Gewolb IH, Panigrahi P. Effects of oral Lactobacillus GG on enteric microflora in low-birth-weight neonates. J Pediatr Gastroenterol Nutr. 2003 Mar;36(3):397-402. doi: 10.1097/00005176-200303000-00019. PMID 12604982
- [Background] Kitajima H, Sumida Y, Tanaka R, Yuki N, Takayama H, Fujimura M. Early administration of Bifidobacterium breve to preterm infants: randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 1997 Mar;76(2):F101-7. doi: 10.1136/fn.76.2.f101. PMID 9135288
- [Background] Caplan MS, Jilling T. Neonatal necrotizing enterocolitis: possible role of probiotic supplementation. J Pediatr Gastroenterol Nutr. 2000;30 Suppl 2:S18-22. No abstract available. PMID 10749397
- [Background] Costalos C, Skouteri V, Gounaris A, Sevastiadou S, Triandafilidou A, Ekonomidou C, Kontaxaki F, Petrochilou V. Enteral feeding of premature infants with Saccharomyces boulardii. Early Hum Dev. 2003 Nov;74(2):89-96. doi: 10.1016/s0378-3782(03)00090-2. PMID 14580749
- [Background] Hoyos AB. Reduced incidence of necrotizing enterocolitis associated with enteral administration of Lactobacillus acidophilus and Bifidobacterium infantis to neonates in an intensive care unit. Int J Infect Dis. 1999 Summer;3(4):197-202. doi: 10.1016/s1201-9712(99)90024-3. PMID 10575148
- [Background] Lin HC, Su BH, Chen AC, Lin TW, Tsai CH, Yeh TF, Oh W. Oral probiotics reduce the incidence and severity of necrotizing enterocolitis in very low birth weight infants. Pediatrics. 2005 Jan;115(1):1-4. doi: 10.1542/peds.2004-1463. PMID 15629973
- [Background] Bin-Nun A, Bromiker R, Wilschanski M, Kaplan M, Rudensky B, Caplan M, Hammerman C. Oral probiotics prevent necrotizing enterocolitis in very low birth weight neonates. J Pediatr. 2005 Aug;147(2):192-6. doi: 10.1016/j.jpeds.2005.03.054. PMID 16126048
- [Background] Deshpande G, Rao S, Patole S. Probiotics for prevention of necrotising enterocolitis in preterm neonates with very low birthweight: a systematic review of randomised controlled trials. Lancet. 2007 May 12;369(9573):1614-20. doi: 10.1016/S0140-6736(07)60748-X. PMID 17499603
- [Background] Salminen S, von Wright A, Morelli L, Marteau P, Brassart D, de Vos WM, Fonden R, Saxelin M, Collins K, Mogensen G, Birkeland SE, Mattila-Sandholm T. Demonstration of safety of probiotics -- a review. Int J Food Microbiol. 1998 Oct 20;44(1-2):93-106. doi: 10.1016/s0168-1605(98)00128-7. PMID 9849787
- [Background] Agostoni C, Axelsson I, Goulet O, Koletzko B, Michaelsen KF, Puntis JW, Rigo J, Shamir R, Szajewska H, Turck D; ESPGHAN Committee on Nutrition. Prebiotic oligosaccharides in dietetic products for infants: a commentary by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2004 Nov;39(5):465-73. doi: 10.1097/00005176-200411000-00003. PMID 15572882
- [Background] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Background] Macfarlane S, Macfarlane GT, Cummings JH. Review article: prebiotics in the gastrointestinal tract. Aliment Pharmacol Ther. 2006 Sep 1;24(5):701-14. doi: 10.1111/j.1365-2036.2006.03042.x. PMID 16918875
- [Background] Moro G, Minoli I, Mosca M, Fanaro S, Jelinek J, Stahl B, Boehm G. Dosage-related bifidogenic effects of galacto- and fructooligosaccharides in formula-fed term infants. J Pediatr Gastroenterol Nutr. 2002 Mar;34(3):291-5. doi: 10.1097/00005176-200203000-00014. PMID 11964956
- [Background] Boehm G, Lidestri M, Casetta P, Jelinek J, Negretti F, Stahl B, Marini A. Supplementation of a bovine milk formula with an oligosaccharide mixture increases counts of faecal bifidobacteria in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2002 May;86(3):F178-81. doi: 10.1136/fn.86.3.f178. PMID 11978748
- [Background] Lidestri M, Agosti M, Marini A, Boehm G. Oligosaccharides might stimulate calcium absorption in formula-fed preterm infants. Acta Paediatr Suppl. 2003 Sep;91(441):91-2. doi: 10.1111/j.1651-2227.2003.tb00654.x. PMID 14599050
- [Background] Knol J, Scholtens P, Kafka C, Steenbakkers J, Gro S, Helm K, Klarczyk M, Schopfer H, Bockler HM, Wells J. Colon microflora in infants fed formula with galacto- and fructo-oligosaccharides: more like breast-fed infants. J Pediatr Gastroenterol Nutr. 2005 Jan;40(1):36-42. doi: 10.1097/00005176-200501000-00007. PMID 15625424
- [Background] Mihatsch WA, Hoegel J, Pohlandt F. Prebiotic oligosaccharides reduce stool viscosity and accelerate gastrointestinal transport in preterm infants. Acta Paediatr. 2006 Jul;95(7):843-8. doi: 10.1080/08035250500486652. PMID 16801182
- [Background] Knol J, Boehm G, Lidestri M, Negretti F, Jelinek J, Agosti M, Stahl B, Marini A, Mosca F. Increase of faecal bifidobacteria due to dietary oligosaccharides induces a reduction of clinically relevant pathogen germs in the faeces of formula-fed preterm infants. Acta Paediatr Suppl. 2005 Oct;94(449):31-3. doi: 10.1111/j.1651-2227.2005.tb02152.x. PMID 16214763
- [Background] Moro G, Arslanoglu S, Stahl B, Jelinek J, Wahn U, Boehm G. A mixture of prebiotic oligosaccharides reduces the incidence of atopic dermatitis during the first six months of age. Arch Dis Child. 2006 Oct;91(10):814-9. doi: 10.1136/adc.2006.098251. Epub 2006 Jul 27. PMID 16873437
- [Background] Szilagyi A. Redefining lactose as a conditional prebiotic. Can J Gastroenterol. 2004 Mar;18(3):163-7. doi: 10.1155/2004/350732. PMID 15054489
- [Background] Schumann C. Medical, nutritional and technological properties of lactulose. An update. Eur J Nutr. 2002 Nov;41 Suppl 1:I17-25. doi: 10.1007/s00394-002-1103-6. PMID 12420112
- [Background] PETUELY F. [Lactobacillus bifidus flora produced in artificially-fed infants by bifidogenic substances (bifidus factor)]. Z Kinderheilkd. 1957;79(2):174-9. No abstract available. German. PMID 13531346
- [Background] Uhlemann M, Heine W, Mohr C, Plath C, Pap S. [Effects of oral administration of bifidobacteria on intestinal microflora in premature and newborn infants]. Z Geburtshilfe Neonatol. 1999 Sep-Oct;203(5):213-7. German. PMID 10596415
- [Background] MACGILLIVRAY PC, FINLAY HV, BINNS TB. Use of lactulose to create a preponderance of Lactobacilli in the intestine of bottle-fed infants. Scott Med J. 1959 Apr;4(4):182-9. doi: 10.1177/003693305900400405. No abstract available. PMID 13646664